CLINICAL TRIAL: NCT00003346
Title: Phase I-II Trial of High-Dose Acetaminophen With Carmustine in Patients With Metastatic Melanoma
Brief Title: Combination Chemotherapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-124; CDR0000066323 (Registry Identifier: PDQ (Physician Data Query)); NCI-H98-0014
Record Dates: First submitted 1999-11-01; First posted 2003-04-25 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Acetaminophen; Acetylcysteine; Carmustine

INTERVENTIONS:
Drug: acetaminophen
Drug: acetylcysteine
Drug: carmustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy consisting of acetaminophen plus carmustine in treating patients who have stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) and the optimal biologic dose (OBD) of high-dose acetaminophen when given alone, and the MTD of carmustine when given with acetaminophen at the OBD in patients with metastatic melanoma (Phase I closed to accrual 3/7/2001).
* Determine the dose of acetaminophen that results in maximal depletion of intracellular glutathione in these patients.
* Assess the antitumor activity of high-dose acetaminophen in these patients.
* Assess the toxicity and antitumor activity of carmustine when administered with high-dose acetaminophen in these patients.

OUTLINE: This is a dose-escalation study.

* Phase I: (closed to accrual 3/7/2001) Patients receive a single oral dose of acetaminophen, then acetylcysteine IV over 20 hours, beginning 6-8 hours after the acetaminophen. This treatment is repeated 3 weeks later. On day 1 of the first treatment, patients also receive carmustine IV over 1 hour, before the acetylcysteine. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients each receive escalating doses of acetaminophen to determine the optimal biological dose (OBD). The OBD is defined as the lowest dose at or preceding the maximum tolerated dose (MTD) that results in maximal depletion of glutathione. The MTD is defined as the dose at which no more than 1 to 6 patients experience dose-limiting toxicity (DLT).

Once the OBD is established for acetaminophen, cohorts of 3-6 patients each receive escalating doses of carmustine. The MTD is defined as for acetaminophen. Dose escalation does not proceed until all patients are observed for 6 weeks after receiving carmustine.

Once the OBD for acetaminophen and MTD for carmustine are determined, 3 more patients are treated at 3 week intervals instead of 6 weeks. If no DLT is observed, this is the dose and schedule for the phase II portion of the study.

* Phase II: A cohort of 14 patients receives oral acetaminophen and acetylcysteine IV every 3 weeks. Another cohort of 14 patients receives oral acetaminophen and acetylcysteine IV, then oral acetaminophen, carmustine IV, and acetylcysteine IV 3 weeks later. Patients continue therapy in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 30-80 patients will be accrued for this study within 40 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV melanoma or stage III melanoma not potentially curable by surgery
* Phase I: (closed to accrual 3/7/2001) measurable or evaluable disease required
* Phase II: At least 2 measurable subcutaneous or cutaneous metastases that are accessible for biopsy

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Hemoglobin at least 9 g/dL
* Platelet count at least 100,000/mm^3
* No active bleeding

Hepatic:

* AST less than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 1.5 times ULN
* PT/PTT within normal range

Renal:

* Not specified

Pulmonary:

* No interstitial lung disease or unexplained interstitial infiltrates on chest x-ray
* No chronic obstructive pulmonary disease
* No asthma requiring treatment

Other:

* No active infection requiring antimicrobial drugs
* Not pregnant or nursing
* Fertile patients must use effective barrier contraception
* No allergies to acetaminophen or acetylcysteine

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin)
* No prior nitrosoureas
* No prior hepatic perfusions with chemotherapy

Endocrine therapy:

* No concurrent oral contraceptives

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* No concurrent vitamin, mineral, or garlic supplements
* At least 7 days since prior garlic or alcohol
* No concurrent treatment with medications known to affect P450 hepatic enzymes
* No concurrent treatment with calcium channel blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 1997-11; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B. Chapman, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States